CLINICAL TRIAL: NCT02730052
Title: Estudio RioplateNsE Sobre Telemonitoreo en hIpertensos No-controlAdos
Brief Title: Telemonitoring of Uncontrolled Hypertension
Acronym: ERNESTINA
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Centers recruited poorly
Sponsor: Universidad de la Republica (Other)
Collaborators: Hospital Italiano de Buenos Aires (Other); KU Leuven (Other)
Responsible Party: Principal Investigator, José Boggia, MD PhD, Universidad de la Republica
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11/16
Record Dates: First submitted 2016-02-28; First posted 2016-04-06 (Estimated); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Hypertension
Keywords: Blood pressure control; Hypertension; Office blood pressure; Self-measured blood pressure,; Telemonitoring
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Omron 9200T without Telemonitoring (Active Comparator): In the control group doctors will receive information on the self-measured blood pressure as recorded at home via a diary card.
  Interventions: Device: Omron 9200T without Telemonitoring
- Omron 9200T plus Telemonitoring (Experimental): In the intervention group, doctors will receive weekly reports via telemonitoring of self-measured blood pressure.
  Interventions: Device: Omron 9200T plus Telemonitoring

INTERVENTIONS:
Device: Omron 9200T plus Telemonitoring — Telemonitoring of the self-measured blood pressure at home. After each blood pressure measurement the values are transmitted to and stored into a central station where a condensed weekly report is elaborated and delivered to the doctor (investigator).
  Other Names: Telemonitored Self-BP Measurement
  Arms: Omron 9200T plus Telemonitoring
Device: Omron 9200T without Telemonitoring — Self-measured blood pressure at home and register the values in a diary card. Participants will perform 2 consecutive blood pressure measurements twice a day for a 7 day period, previous to the visit to the doctor's (investigator) office.
  Other Names: Conventional Self-BP Measurement
  Arms: Omron 9200T without Telemonitoring

SUMMARY:
The proportion of hypertensive patients achieving adequate blood pressure control meeting guideline targets remains low. Of those patients on blood pressure lowering drugs, only 50% reach control.

Objectives:

1. Test the feasibility of telemonitoring of blood pressure in uncontrolled hypertensive patients.
2. Investigate whether telemonitoring enabled self-measurement of blood pressure leads to faster blood pressure control than self-measurement without telemonitoring.
3. Secondary endpoints include adverse effects, assessment of quality of life, adherence, a log of technical problems, and cost-effectiveness.

Methods:

Randomised parallel-group study consisting of 4 stages.

* Screening to check for eligibility.
* Randomisation in a 1:1 proportion to control or experimental arm: In the control arm, doctors will receive reports on the self-measured blood pressure based on diary cards; in the experimental group, doctors will receive weekly reports via telemonitoring.
* Treatment period: Doctors will adjust treatment according to the present guidelines of Hypertension. Blood pressure control is a home blood pressure below 135 mm Hg systolic and 85 mm Hg diastolic. Once blood pressure control is achieved the treatment period ends.
* Late follow-up: Assessment of blood pressure control at home 3 months after completion of the treatment period by means of telemonitoring.

Sample size: 120 patients per group. Patients: recruited at clinics from Uruguay and Argentina.

Main Inclusion Criteria:

* Women and men, age range 20 to 80 years.
* Uncontrolled hypertension and new diagnosed hypertension with a self-measured blood pressure at home of 135 mm Hg systolic and/or 85 mm Hg diastolic or more;
* Patients should be willing to accept adherence checking during follow-up and sign an informed written consent.

Exclusion Criteria

* Patients emotionally or intellectually not capable of measuring their blood pressure at home;
* A clinical or social context, which is suboptimal for the self-measurement of blood pressure;
* Pregnancy;
* Alcohol or substance abuse or psychiatric illnesses;
* Participation in another study. Expected outcomes: blood pressure control will be achieved faster in the telemonitoring group.

DETAILED DESCRIPTION:
1. Research Questions

   Previous studies demonstrated the feasibility of telemonitoring of blood pressure. However, several issues remain unaddressed.
   * Feasibility of telemonitoring within the South American context has never been tested. No attempt has ever been made in South America to assess adherence to antihypertensive drugs in primary care.
   * Telemonitoring of blood pressure will never make it to the routine clinical practice unless it can be proven that application of the technique results in faster and better blood pressure control compared with usual care including self-measurement of blood pressure at home.
   * Secondary endpoints must also include adverse events, a simple assessment of quality of life, adherence, a log of technical problems, and cost-effectiveness.
2. General Design

   ERNESTINA is a randomised parallel-group study, which will address the feasibility and potential benefits of telemonitoring of blood pressure at home. Eligible patients will be recruited at outpatient medical clinics.

   - Screening period followed by stratification and randomisation: Screening involves checking inclusion and exclusion criteria, ruling out secondary hypertension remediable by specific treatment, and obtaining informed written consent as outlined in the Helsinki declaration.

   Eligible patients will be stratified by centre and randomised in a one-to-one proportion to control or intervention. Randomisation will be implemented by sequentially numbered sealed envelopes, which contain the group assignment. These envelopes will be available at the practices, so that no contact with the Studies Coordinating Centre (SCC) will be necessary to randomise the patient.

   - Randomised period: Investigators will optimise medical treatment by rotating patients through different classes of antihypertensive drugs, combining drug classes according to the current guidelines of the Argentinian and European Societies of Hypertension (SAHA and ESH), while achieving the maximal tolerated dose of each drug. In the intervention group, investigators will receive a report on the telemonitoring data at weekly intervals; in the control group doctors will receive information on the self-measured blood pressure as recorded at home in the week preceding the office visit via a diary card. Doctors are free to schedule contacts with their patients and office visits at their own discretion but visits should be at least every 3 weeks. Once blood pressure control is achieved, the blood pressure measuring devices (telemonitoring enabled or not) will be recuperated and will become available for a next patient. In the control group, patients will keep a diary card in the week preceding the office visits.

   - Late follow-up: Three months after achieving blood pressure control, all patients will be telemonitored for 1 week and complete a diary card, preceding an office visit.
3. Primary and Secondary Endpoints

Primary endpoint

The primary endpoint will be the time to blood pressure control in the two randomised groups. Blood pressure control will be defined as a self-measured blood pressure at home below 135 mm Hg systolic and 85 mm Hg diastolic. Blood pressure control is assumed to be present if the aforementioned levels are attained during the week preceding the last office visit of the randomised treatment visit. Treatment resistance is a home blood pressure not controlled on 3 drugs classes given at maximal doses, preferably including a diuretic after 6 months of follow-up. These patients might be referred for further exploration and treatment adjustment to a hypertension centre.

Secondary endpoints

Secondary endpoints related to blood pressure control (efficacy) are:

* The proportion of patients reaching blood pressure control on self-measurement at home and office measurement; Blood pressure control on office measurement is a seated blood pressure below 140 mm Hg systolic and 90 mm Hg;
* The proportion of patients reaching and maintaining blood pressure control on self-measurement and office measurement at the late follow-up visit;
* The intensity of medical treatment;
* Adverse events, recorded by a self-administered questionnaire.
* Assessment of drug adherence;
* Assessment of quality of life;
* Analysis of cost-effectiveness.

Economic Analysis The cost-effectiveness analysis will include both the direct and indirect costs of the intervention. The costs will be balanced against the use of medical resources, including visits, medications, and use of medical resources.

Moreover, the incremental cost-effectiveness ratios (ICERs) will be calculated by dividing the net cost of intervention by the total incremental health care costs after the intervention according to the formula ICER = (Ci - Cc) / (Ei - Ec), where Ci and Cc and Ei and Ec are the costs and effectiveness associated with the intervention and usual care, respectively. Sensitivity analyses will examine the influence of uncertainty in the variables and assumptions. Model performance will be estimated through confidence intervals estimated in a probabilistic manner using Monte Carlo simulation.

ELIGIBILITY:
Inclusion Criteria:

1. Women and men are eligible. Women of reproductive age should apply effective contraception.
2. Age ranges from 20 years (inclusive) to 80 years.
3. At screening, patients should have hypertension, which is uncontrolled on medical treatment. Uncontrolled hypertension is an office blood pressure of 140 mm Hg systolic or 90 mm Hg diastolic or higher AND a self-measured blood pressure at home of 135 mm Hg systolic or 85 mm Hg diastolic or more. Practitioners will receive a weekly report on the self-measured blood pressure at home summarising the results of the run-in period.
4. At the screening visit, patients should either be untreated for at least 4 weeks or taking a stable drug regimen for at least 4 weeks. Medical treatment can consist of all major drug classes. This includes diuretics, beta-blockers, alfa-blockers, calcium-channel blockers (CCBs), inhibitors of the renin system (angiotensin-converting enzyme inhibitors (ACEIs), angiotensin II type 1 receptor blockers (ARBs), the direct renin inhibitor aliskiren,18 aldosterone receptor antagonists (ARAs), centrally acting antihypertensive drugs and vasodilators (hydralazine). In line with current recommendations and recent studies, unless contra-indicated or not tolerated, aldosterone antagonists, such as spironolactone 25 to 50 mg per day should have been attempted for at least 4 weeks to improve blood pressure control in treatment-resistant patients. (1) The patients should be intellectually and emotionally capable of measuring their blood pressure at home and accept to keep a diary (control group) or to have a report sent to their doctor (intervention group).
5. Patient should provide written informed consent.

Exclusion Criteria:

1. The clinical context is suboptimal for telemonitoring of blood pressure:

   * Myocardial infarction, unstable angina pectoris, or a cerebrovascular accident within 6 months of the screening period;
   * Type 1 diabetes mellitus requiring multiple adjustments of treatment to maintain control or diabetes mellitus with recent hyperglycaemic or hypoglycaemic coma;
   * Renal dysfunction defined as an estimated glomerular filtration rate (eGFR) of less than 30 mL/min/1.73m2, using the Modification of Diet in Renal Disease formula;
   * Secondary hypertension, in which treatment options other than antihypertensive drug treatment are indicated;
   * Sleep apnea syndrome that qualifies for treatment with continuous positive airway pressure (CPAP);
   * Atrial fibrillation or arrhythmia making oscillometric blood pressure measurement unreliable;
   * The patient is on a waiting list for elective surgery or a cardiovascular intervention;
   * Patients with alcohol or substance abuse or psychiatric illnesses.
2. The patients should not have any serious medical condition, which in the opinion of the investigator, may adversely interfere with self-measurement of blood pressure at home.
3. Patients should not participate in any other trial of an investigational drug or device.

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-12; Primary Completion 2019-06 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Time to blood pressure control | through study completion, an average of 2 years
  Blood pressure control will be defined as a self-measured blood pressure at home below 135 mm Hg systolic and 85 mm Hg diastolic. Blood pressure control is assumed to be present if the aforementioned levels are attained during the preceding week to medical control.

SECONDARY OUTCOMES:
The proportion of patients reaching blood pressure control on self-measurement at home and office measurement | through study completion, an average of 2 years
  For each participant, the individual time frame is up-to 6 months. However, to know the proportion of patients we need to recruit at least 50% of the calculated sample.
  Blood pressure control on office measurement is an average (3 consecutive readings) blood pressure below 140 mm Hg systolic and 90 mm Hg.
  Blood pressure control on self-blood pressure measurement is an average (up to 28 readings) blood pressure below 135 mm Hg systolic and 85 mm Hg diastolic.
The proportion of patients reaching and maintaining blood pressure control on self-measurement and office measurement at the late follow-up visit | through study completion, an average of 2 years
  For each participant, the individual time frame is up-to 6 months. However, to know the proportion of patients we need to recruit at least 50% of the calculated sample.
  Blood pressure control on office measurement is an average (3 consecutive readings) blood pressure below 140 mm Hg systolic and 90 mm Hg.
  Blood pressure control on self-blood pressure measurement is an average (up to 28 readings) blood pressure below 135 mm Hg systolic and 85 mm Hg diastolic.
Total pill load per day | through study completion, an average of 2 years
  For each participant, the individual time frame is up-to 6 months. However, to know the proportion of patients we need to recruit at least 50% of the calculated sample.
  We will compute total pill load per day and number of single-pill combinations of anti-hypertensive medication at the moment of reaching blood pressure control or leaving the study.
Number of single-pill combinations | through study completion, an average of 2 years
  For each participant, the individual time frame is up-to 6 months. However, to know the proportion of patients we need to recruit at least 50% of the calculated sample.
  We will compute total pill load per day and number of single-pill combinations of anti-hypertensive medication at the moment of reaching blood pressure control or leaving the study.
Adverse events, recorded by a self-administered questionnaire | through study completion, an average of 2 years
  For each participant, the individual time frame is up-to 6 months. However, to know the proportion of patients we need to recruit at least 50% of the calculated sample.
Assessment of drug adherence using Morisky questionnaire | through study completion, an average of 2 years
  We will use Morisky questionaire to asses adherence to anti-hypertensive treatment
Assessment of quality of life using the Euro-Quality-of-life questionnaire "EQ-5D-5L" | through study completion, an average of 2 years
Health care costs from randomization to last follow-up | through study completion, an average of 2 years
  For each participant, the individual time frame is up-to 6 months. However, to know the proportion of patients we need to recruit at least 50% of the calculated sample.
  Cost will include both the direct and indirect costs of the intervention. The costs will be balanced against the use of medical resources, including visits, medications, and use of medical resources. The incremental cost-effectiveness ratios (ICERs) will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Jose G Boggia, MD PhD, Principal Investigator — Universidad de la Republica - Uruguay
Locations (8):
- Argentina (4):
  - Center AR-4, Córdoba, Córdoba Province
  - Center AR-3, Rosario, Santa Fe Province
  - Center AR-1, Buenos Aires
  - Center AR-2, Buenos Aires
- Uruguay (4):
  - Center UY-1, Montevideo
  - Center UY-2, Montevideo
  - Center UY-3, Montevideo
  - Center UY-4, Montevideo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aparicio LS, Thijs L, Boggia J, Jacobs L, Barochiner J, Odili AN, Alfie J, Asayama K, Cuffaro PE, Nomura K, Ohkubo T, Tsuji I, Stergiou GS, Kikuya M, Imai Y, Waisman GD, Staessen JA; International Database on Home Blood Pressure in Relation to Cardiovascular Outcome (IDHOCO) Investigators. Defining thresholds for home blood pressure monitoring in octogenarians. Hypertension. 2015 Oct;66(4):865-73. doi: 10.1161/HYPERTENSIONAHA.115.05800. Epub 2015 Jul 27. PMID 26355122
- [Background] Staessen JA, Kuznetsova T, Stolarz K. Hypertension prevalence and stroke mortality across populations. JAMA. 2003 May 14;289(18):2420-2. doi: 10.1001/jama.289.18.2420. No abstract available. PMID 12746368
- [Background] Weinehall L, Ohgren B, Persson M, Stegmayr B, Boman K, Hallmans G, Lindholm LH. High remaining risk in poorly treated hypertension: the 'rule of halves' still exists. J Hypertens. 2002 Oct;20(10):2081-8. doi: 10.1097/00004872-200210000-00029. PMID 12359988
- [Background] Burnier M. Medication adherence and persistence as the cornerstone of effective antihypertensive therapy. Am J Hypertens. 2006 Nov;19(11):1190-6. doi: 10.1016/j.amjhyper.2006.04.006. PMID 17070434
- [Background] Calhoun DA, Jones D, Textor S, Goff DC, Murphy TP, Toto RD, White A, Cushman WC, White W, Sica D, Ferdinand K, Giles TD, Falkner B, Carey RM; American Heart Association Professional Education Committee. Resistant hypertension: diagnosis, evaluation, and treatment: a scientific statement from the American Heart Association Professional Education Committee of the Council for High Blood Pressure Research. Circulation. 2008 Jun 24;117(25):e510-26. doi: 10.1161/CIRCULATIONAHA.108.189141. PMID 18574054
- [Background] Pickering TG. Home blood pressure monitoring: a new standard method for monitoring hypertension control in treated patients. Nat Clin Pract Cardiovasc Med. 2008 Dec;5(12):762-3. doi: 10.1038/ncpcardio1374. Epub 2008 Oct 14. PMID 18852711
- [Background] Parati G, Omboni S, Albini F, Piantoni L, Giuliano A, Revera M, Illyes M, Mancia G; TeleBPCare Study Group. Home blood pressure telemonitoring improves hypertension control in general practice. The TeleBPCare study. J Hypertens. 2009 Jan;27(1):198-203. doi: 10.1097/hjh.0b013e3283163caf. PMID 19145785
- [Background] Logan AG, Irvine MJ, McIsaac WJ, Tisler A, Rossos PG, Easty A, Feig DS, Cafazzo JA. Effect of home blood pressure telemonitoring with self-care support on uncontrolled systolic hypertension in diabetics. Hypertension. 2012 Jul;60(1):51-7. doi: 10.1161/HYPERTENSIONAHA.111.188409. Epub 2012 May 21. PMID 22615116
- [Background] McCant F, McKoy G, Grubber J, Olsen MK, Oddone E, Powers B, Bosworth HB. Feasibility of blood pressure telemonitoring in patients with poor blood pressure control. J Telemed Telecare. 2009;15(6):281-5. doi: 10.1258/jtt.2009.090202. PMID 19720764
- [Background] Bosworth HB, Olsen MK, Dudley T, Orr M, Goldstein MK, Datta SK, McCant F, Gentry P, Simel DL, Oddone EZ. Patient education and provider decision support to control blood pressure in primary care: a cluster randomized trial. Am Heart J. 2009 Mar;157(3):450-6. doi: 10.1016/j.ahj.2008.11.003. Epub 2009 Jan 10. PMID 19249414
- [Background] Bosworth HB, Olsen MK, McCant F, Harrelson M, Gentry P, Rose C, Goldstein MK, Hoffman BB, Powers B, Oddone EZ. Hypertension Intervention Nurse Telemedicine Study (HINTS): testing a multifactorial tailored behavioral/educational and a medication management intervention for blood pressure control. Am Heart J. 2007 Jun;153(6):918-24. doi: 10.1016/j.ahj.2007.03.004. PMID 17540191
- [Background] Bosworth HB, Powers BJ, Olsen MK, McCant F, Grubber J, Smith V, Gentry PW, Rose C, Van Houtven C, Wang V, Goldstein MK, Oddone EZ. Home blood pressure management and improved blood pressure control: results from a randomized controlled trial. Arch Intern Med. 2011 Jul 11;171(13):1173-80. doi: 10.1001/archinternmed.2011.276. PMID 21747013
- [Background] 41st World Medical Assembly. Declaration of Helsinki : recommendations guiding physicians in biomedical research involving human subjects. Bull Pan Am Health Organ 1990; 24: 606-609
- [Background] Mancia G, Fagard R, Narkiewicz K, Redon J, Zanchetti A, Bohm M, Christiaens T, Cifkova R, De Backer G, Dominiczak A, Galderisi M, Grobbee DE, Jaarsma T, Kirchhof P, Kjeldsen SE, Laurent S, Manolis AJ, Nilsson PM, Ruilope LM, Schmieder RE, Sirnes PA, Sleight P, Viigimaa M, Waeber B, Zannad F; Task Force Members. 2013 ESH/ESC Guidelines for the management of arterial hypertension: the Task Force for the management of arterial hypertension of the European Society of Hypertension (ESH) and of the European Society of Cardiology (ESC). J Hypertens. 2013 Jul;31(7):1281-357. doi: 10.1097/01.hjh.0000431740.32696.cc. No abstract available. PMID 23817082
- [Background] Staessen JA, Byttebier G, Buntinx F, Celis H, O'Brien ET, Fagard R. Antihypertensive treatment based on conventional or ambulatory blood pressure measurement. A randomized controlled trial. Ambulatory Blood Pressure Monitoring and Treatment of Hypertension Investigators. JAMA. 1997 Oct 1;278(13):1065-72. PMID 9315764
- [Background] Staessen JA, Den Hond E, Celis H, Fagard R, Keary L, Vandenhoven G, O'Brien ET; Treatment of Hypertension Based on Home or Office Blood Pressure (THOP) Trial Investigators. Antihypertensive treatment based on blood pressure measurement at home or in the physician's office: a randomized controlled trial. JAMA. 2004 Feb 25;291(8):955-64. doi: 10.1001/jama.291.8.955. PMID 14982911
- [Background] Briggs AH. Handling uncertainty in cost-effectiveness models. Pharmacoeconomics. 2000 May;17(5):479-500. doi: 10.2165/00019053-200017050-00006. PMID 10977389
- [Background] Staessen JA, Li Y, Richart T. Oral renin inhibitors. Lancet. 2006 Oct 21;368(9545):1449-56. doi: 10.1016/S0140-6736(06)69442-7. PMID 17055947
- [Background] Calhoun DA, White WB. Effectiveness of the selective aldosterone blocker, eplerenone, in patients with resistant hypertension. J Am Soc Hypertens. 2008 Nov-Dec;2(6):462-8. doi: 10.1016/j.jash.2008.05.005. Epub 2008 Jul 23. PMID 20409927
- [Background] Levey AS, Bosch JP, Lewis JB, Greene T, Rogers N, Roth D. A more accurate method to estimate glomerular filtration rate from serum creatinine: a new prediction equation. Modification of Diet in Renal Disease Study Group. Ann Intern Med. 1999 Mar 16;130(6):461-70. doi: 10.7326/0003-4819-130-6-199903160-00002. PMID 10075613
- [Background] Levey AS, Stevens LA, Schmid CH, Zhang YL, Castro AF 3rd, Feldman HI, Kusek JW, Eggers P, Van Lente F, Greene T, Coresh J; CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration). A new equation to estimate glomerular filtration rate. Ann Intern Med. 2009 May 5;150(9):604-12. doi: 10.7326/0003-4819-150-9-200905050-00006. PMID 19414839
- [Background] Consensus statement on the definition of orthostatic hypotension, pure autonomic failure, and multiple system atrophy. The Consensus Committee of the American Autonomic Society and the American Academy of Neurology. Neurology. 1996 May;46(5):1470. doi: 10.1212/wnl.46.5.1470. No abstract available. PMID 8628505
- [Background] Expert Committee on the Diagnosis and Classification of Diabetes Mellitus. Report of the expert committee on the diagnosis and classification of diabetes mellitus. Diabetes Care. 2003 Jan;26 Suppl 1:S5-20. doi: 10.2337/diacare.26.2007.s5. No abstract available. PMID 12502614
- [Background] British Cardiac Society; British Hypertension Society; Diabetes UK; HEART UK; Primary Care Cardiovascular Society; Stroke Association. JBS 2: Joint British Societies' guidelines on prevention of cardiovascular disease in clinical practice. Heart. 2005 Dec;91 Suppl 5(Suppl 5):v1-52. doi: 10.1136/hrt.2005.079988. No abstract available. PMID 16365341
- [Background] Chobanian AV, Bakris GL, Black HR, Cushman WC, Green LA, Izzo JL Jr, Jones DW, Materson BJ, Oparil S, Wright JT Jr, Roccella EJ; Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure. National Heart, Lung, and Blood Institute; National High Blood Pressure Education Program Coordinating Committee. Seventh report of the Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure. Hypertension. 2003 Dec;42(6):1206-52. doi: 10.1161/01.HYP.0000107251.49515.c2. Epub 2003 Dec 1. PMID 14656957
- [Background] Pimenta E, Gaddam KK, Oparil S, Aban I, Husain S, Dell'Italia LJ, Calhoun DA. Effects of dietary sodium reduction on blood pressure in subjects with resistant hypertension: results from a randomized trial. Hypertension. 2009 Sep;54(3):475-81. doi: 10.1161/HYPERTENSIONAHA.109.131235. Epub 2009 Jul 20. PMID 19620517
- [Background] Claxton AJ, Cramer J, Pierce C. A systematic review of the associations between dose regimens and medication compliance. Clin Ther. 2001 Aug;23(8):1296-310. doi: 10.1016/s0149-2918(01)80109-0. PMID 11558866
- [Background] Chapman RH, Benner JS, Petrilla AA, Tierce JC, Collins SR, Battleman DS, Schwartz JS. Predictors of adherence with antihypertensive and lipid-lowering therapy. Arch Intern Med. 2005 May 23;165(10):1147-52. doi: 10.1001/archinte.165.10.1147. PMID 15911728
- [Background] Hernandez-Hernandez R, Armas de Hernandez MJ, Armas-Padilla MC, Carvajal AR, Guerrero-Pajuelo J. The effects of missing a dose of enalapril versus amlodipine on ambulatory blood pressure. Blood Press Monit. 1996 Apr;1(2):121-126. PMID 10226213
- [Background] Lowy A, Munk VC, Ong SH, Burnier M, Vrijens B, Tousset EP, Urquhart J. Effects on blood pressure and cardiovascular risk of variations in patients' adherence to prescribed antihypertensive drugs: role of duration of drug action. Int J Clin Pract. 2011 Jan;65(1):41-53. doi: 10.1111/j.1742-1241.2010.02569.x. Epub 2010 Nov 22. PMID 21091596
- [Background] Staessen JA, Fagard R, Thijs L, Celis H, Arabidze GG, Birkenhager WH, Bulpitt CJ, de Leeuw PW, Dollery CT, Fletcher AE, Forette F, Leonetti G, Nachev C, O'Brien ET, Rosenfeld J, Rodicio JL, Tuomilehto J, Zanchetti A. Randomised double-blind comparison of placebo and active treatment for older patients with isolated systolic hypertension. The Systolic Hypertension in Europe (Syst-Eur) Trial Investigators. Lancet. 1997 Sep 13;350(9080):757-64. doi: 10.1016/s0140-6736(97)05381-6. PMID 9297994
- [Background] Staessen JA, Wang JG, Brand E, Barlassina C, Birkenhager WH, Herrmann SM, Fagard R, Tizzoni L, Bianchi G. Effects of three candidate genes on prevalence and incidence of hypertension in a Caucasian population. J Hypertens. 2001 Aug;19(8):1349-58. doi: 10.1097/00004872-200108000-00002. PMID 11518842
- [Background] Stolarz-Skrzypek K, Kuznetsova T, Thijs L, Tikhonoff V, Seidlerova J, Richart T, Jin Y, Olszanecka A, Malyutina S, Casiglia E, Filipovsky J, Kawecka-Jaszcz K, Nikitin Y, Staessen JA; European Project on Genes in Hypertension (EPOGH) Investigators. Fatal and nonfatal outcomes, incidence of hypertension, and blood pressure changes in relation to urinary sodium excretion. JAMA. 2011 May 4;305(17):1777-85. doi: 10.1001/jama.2011.574. PMID 21540421
- [Background] Boggia J, Thijs L, Hansen TW, Li Y, Kikuya M, Bjorklund-Bodegard K, Richart T, Ohkubo T, Jeppesen J, Torp-Pedersen C, Dolan E, Kuznetsova T, Olszanecka A, Tikhonoff V, Malyutina S, Casiglia E, Nikitin Y, Lind L, Maestre G, Sandoya E, Kawecka-Jaszcz K, Imai Y, Wang J, Ibsen H, O'Brien E, Staessen JA; International Database on Ambulatory blood pressure in relation to Cardiovascular Outcomes Investigators. Ambulatory blood pressure monitoring in 9357 subjects from 11 populations highlights missed opportunities for cardiovascular prevention in women. Hypertension. 2011 Mar;57(3):397-405. doi: 10.1161/HYPERTENSIONAHA.110.156828. Epub 2011 Jan 24. PMID 21263119
- [Background] Beckett NS, Peters R, Fletcher AE, Staessen JA, Liu L, Dumitrascu D, Stoyanovsky V, Antikainen RL, Nikitin Y, Anderson C, Belhani A, Forette F, Rajkumar C, Thijs L, Banya W, Bulpitt CJ; HYVET Study Group. Treatment of hypertension in patients 80 years of age or older. N Engl J Med. 2008 May 1;358(18):1887-98. doi: 10.1056/NEJMoa0801369. Epub 2008 Mar 31. PMID 18378519
- [Background] Haller H, Ito S, Izzo JL Jr, Januszewicz A, Katayama S, Menne J, Mimran A, Rabelink TJ, Ritz E, Ruilope LM, Rump LC, Viberti G; ROADMAP Trial Investigators. Olmesartan for the delay or prevention of microalbuminuria in type 2 diabetes. N Engl J Med. 2011 Mar 10;364(10):907-17. doi: 10.1056/NEJMoa1007994. PMID 21388309
- [Background] Nyholt DR. Genetic case-control association studies--correcting for multiple testing. Hum Genet. 2001 Nov;109(5):564-7. doi: 10.1007/s00439-001-0611-4. Epub 2001 Oct 19. No abstract available. PMID 11735033